CLINICAL TRIAL: NCT05121896
Title: Investigating Neural Plasticity and Nuclear Hyperexcitability in Patients With Oral-ocular Facial Synkinesis Using 7 Tesla Functional MRI
Brief Title: Functional MRI Study Facial Synkinesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL78991.068.21
Record Dates: First submitted 2021-11-02; First posted 2021-11-16 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Facial Synkinesis
Keywords: functional MRI (fMRI); Neural plasticity; Nuclear hyperexcitability
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with facial synkinesis (Active Comparator): Functional MRI scan of the primary and secondary somatosensory cortexes, the primary motor cortex, the supplementary motor cortex, and the ventral lateral premotor cortex while the participant performs motor and sensory tasks.
  Interventions: Device: MRI Scan
- Control participants (Active Comparator): Functional MRI scan of the primary and secondary somatosensory cortexes, the primary motor cortex, the supplementary motor cortex, and the ventral lateral premotor cortex while the participant performs motor and sensory tasks.
  Interventions: Device: MRI Scan

INTERVENTIONS:
Device: MRI Scan — 7.0 tesla functional MRI scan

SUMMARY:
Rationale. Facial synkinesis is one of the most common consequences after facial paralysis, defined as the inability to move muscles due to nerve damage. Facial synkinesis arises during recovery of nerve injury and is characterized by involuntary and synchronous contractions of muscles during facial movements. Patients' quality of life is major influenced by the disease. As patients experience problems with facial movements, this leads to difficulties in expressing emotions, eating, and drinking.

A common type of facial synkinesis is oral-ocular synkinesis, defined as eye closure during movement with the mouth. During movements of the mouth, the buccinator muscle plays an essential role. Both the trigeminal and the facial nerve innervate the buccinator muscle, resulting in a complex sensorimotor feedback system between the nerves. Dysregulation of this feedback system is assumed to result in hyperexcitability of the trigeminal and facial nuclei in the pons. In addition, this will lead to cortical plasticity of the sensory and motor areas of the brain. Based on this, the investigators hypothesize dysregulation of the sensorimotor feedback system in patients with facial synkinesis, resulting in differences in the neuroplastic organization of the primary and secondary somatosensory cortexes, the primary motor cortex, the supplementary motor cortex, and the ventral lateral premotor cortex compared to healthy control participants. In addition, the investigators expect hyperexcitability of the trigeminal and facial nuclei. Therefore, this study aims to obtain a more detailed understanding of the neural reorganization of the sensory and motor areas as a consequence of facial synkinesis using 7T fMRI.

Objective. To study the neuroplasticity of the brain due to facial synkinesis by assessing the somatotopy of the face on several cortexes of interest (primary and secondary somatosensory cortexes, the primary motor cortex, the supplementary motor cortex, and the ventral lateral premotor cortex) compared to healthy control participants.

Study design. A single center imaging study carried out in MUMC+. Study population. Two patients with severe oral-ocular synkinesis will be included in this pilot study. In addition, two age- and sex-matched healthy control participants will be included.

Intervention. Every subject will undergo a single functional MRI scan in the 7 Tesla MRI scan of Scannexus. A scanning session takes approximately 1 hour. During the scan, participants are asked to perform motor and sensory tasks.

Main study parameters. The main study parameter is the hemodynamic response after stimulation of specific parts of the face. Within the areas of interest (primary motor cortex, the ventral lateral premotor cortex, the supplementary motor cortex, the primary somatosensory cortex (S1), and the secondary somatosensory cortex (S2)), the temporo-spatial brain activity patterns after the different motor and sensory tasks are assessed, and the representation of the face is mapped on the cortexes of interest.

ELIGIBILITY:
Inclusion Criteria for all participants:

* absence of facial nerve transposition;
* participants must be 18 years of age or older;
* signed informed consent.

Inclusion Criteria for patients with facial synkinesis:

* patients must have severe facial synkinesis based on the Sunnybrook facial grading system at the time the MRI scan is performed
* synkinesis must occur only on one side of the face

Exclusion Criteria for all participants:

* previous neurosurgery
* contraindications for MRI investigation, such as a pacemaker, implanted pumps or stimulators, iron materials (e.g., piercings), facial tattoos and permanent make up, or claustrophobia.

Exclusion Criteria for control participants:

* control participants must have no forms of facial paralysis prior to the MRI examination and at the time of the MRI procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The neuroplasticity of the brain after facial synkinesis will be measured using functional MRI | Total MRI scan will take 60 minutes
  Changes in the blood oxygen level dependent (BOLD) contrast as a function of motor and sensory tasks of the face will be measured using fMRI.
hyperexcitability of the pons as a result of synkinesis will be measured using functional MRI | Total MRI scan will take 60 minutes
  hyperexcitability of the pons as a result of oral-ocular facial synkinesis compared to the contralateral side or healthy control participants will be measured using fMRI.

SECONDARY OUTCOMES:
Differences in the somatotopy of the sensory area between patients with oral-ocular facial synkinesis compared to healthy control participants will be mapped using functional MRI. | Total MRI scan will take 60 minutes
  Differences between groups in somatotopy of the face in the somatosensory cortex will be assessed using fMRI.
Differences in the somatotopy of the motor area between patients with oral-ocular facial synkinesis compared to healthy control participants will be mapped using functional MRI. | Total MRI scan will take 60 minutes
  Differences between groups in somatotopy of the face in the motor cortex will be assessed using fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Tuinder, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided